CLINICAL TRIAL: NCT03359395
Title: Effects of Pre-medication With Alfentanil on Hemodynamics During and Immediately Following Electroconvulsive Therapy (ECT)
Brief Title: Pre-medication With Alfentanil vs Placebo During ECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00045800
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2020-02

CONDITIONS: Blood Pressure; Electroconvulsive Therapy
Keywords: Anesthesia
MeSH Terms: interventions — Alfentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: study med prepared by a provider not involved in the anesthesia care of the subject
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alfentanil (Active Comparator)
  Interventions: Drug: Alfentanil
- placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Alfentanil — Administration of alfentanil during the induction and maintenance of anesthesia for electroconvulsive therapy to be performed
  Arms: Alfentanil
Drug: Placebos — Administration of a equidose placebo during the induction and maintenance of anesthesia for electroconvulsive therapy to be performed
  Arms: placebo

SUMMARY:
Hemodynamic changes associated with the conduct of electroconvulsive therapy may be minimized with the administration of alfentanil as part of their anesthetic regimen. This study proposes to compare the effects in a blinded fashion. Currently alfentanil is an FDA approved drug used on a daily basis by anesthesiologists on other surgeries so this is not a new indication.

DETAILED DESCRIPTION:
Electroconvulsive therapy is associated with brief hemodynamic alterations that in some patients may be well outside the range of normalcy and potentially dangerous to the patient (Duma A, et al). This cardiovascular response is caused by activation of the autonomic nervous system and consists of an initial parasympathetic response rapidly followed by sympathetically mediated tachycardia and hypertension. The ultra-short acting synthetic opioid alfentanil has a rapid onset and duration of action that mirrors the duration of hemodynamic perturbation associated with Electroconvulsive Therapy (ECT) while having minimal or no effect on the duration or quality of the seizure. This drug may be effective in blunting the hemodynamic perturbations associated with ECT with a minimal amount of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age > /=18 years
* Males or females
* Anticipating electroconvulsive therapy to treat refractory depressive disorder

Exclusion Criteria:

* Under the age of 18
* Allergy to alfentanil
* Allergy to other standard anesthetic medications utilized in the course of ECT (glycopyrrolate, methohexital, and succinylcholine)
* History of malignant hyperthermia
* History of severe airway obstruction, bronchospasm or laryngospasm
* History of recent myocardial infarction, ventricular arrhythmia
* Adverse reaction to ECT requiring premedication with lidocaine or atropine
* Non-English speaking
* Patients unable to consent for themselves
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quinn McCutchen, MD, Principal Investigator — Wake Forest School of Medicne
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCutchen TM, Gligorovic PV, Tighe NTG, Templeton TW, Saha AK. Alfentanil Pretreatment for Electroconvulsive Therapy-Associated Hemodynamic Lability: A Prospective Randomized Crossover Trial. J ECT. 2023 Jun 1;39(2):84-90. doi: 10.1097/YCT.0000000000000885. Epub 2022 Oct 1. PMID 36215414

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One Subject Withdrew before randomization
Groups:
- Alfentanil Then Placebo: Alfentanil: Administration of alfentanil during the induction and maintenance of anesthesia for electroconvulsive therapy to be performed
- Placebo Then Afentanil: Placebos: Administration of a equidose placebo during the induction and maintenance of anesthesia for electroconvulsive therapy to be performed
Period: First Intervention A / B
Arm/Group | Alfentanil Then Placebo | Placebo Then Afentanil
Started | 49 | 50
Completed | 46 | 47
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 2 | 3
Period: Second Intervention B/A
Arm/Group | Alfentanil Then Placebo | Placebo Then Afentanil
Started | 46 | 47
Completed | 43 | 44
Not Completed | 3 | 3
Not completed — Exclusion criteria | 0 | 1
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Alfentanil Then Placebo Arm 1: Alfentanil: Administration of alfentanil during the induction and maintenance of anesthesia for electroconvulsive therapy to be performed
- Placebo Then Alfentanil Arm 2: Placebos: Administration of a equidose placebo during the induction and maintenance of anesthesia for electroconvulsive therapy to be performed
- Total: Total of all reporting groups
Arm/Group | Alfentanil Then Placebo Arm 1 | Placebo Then Alfentanil Arm 2 | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.34 (17.10) | 51.94 (13.96) | 51.621 (15.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 32 | 67
  Male | 14 | 18 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 48 | 48 | 96
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 48 | 46 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 50 | 99
Height (cm) [Mean (Standard Deviation); unit: Centimeters] | 167.57 (11.31) | 167.59 (10.25) | 167.58 (10.67)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 86.28 (31.57) | 85.156 (27.33) | 85.405 (30.05)

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure Change
Description: comparison of Systolic blood pressure changes alfentanil vs placebo
Time Frame: Baseline and up to 90 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Alfentanil | Placebo
Number analyzed (Participants) | 87 | 87
mmHg | 22.011 (36.968) | 38.908 (33.50864)

2. Secondary Outcome: Diastolic Blood Pressure Change
Description: comparison of diastolic blood pressure change alfentanil vs placebo
Time Frame: Baseline and up to 90 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Alfentanil | Placebo
Number analyzed (Participants) | 87 | 87
mmHg | 15.26 (23.3848507043) | 23.34 (24.40)

3. Secondary Outcome: Heart Rate
Description: comparison of heart rate change alfentanil vs placebo
Time Frame: Baseline and up to 15 seconds
Measure: Mean (Standard Deviation); unit: Beats per Minute
Arm/Group | Alfentanil | Placebo
Number analyzed (Participants) | 87 | 87
Beats per Minute | 26.00 (19.823) | 28.197674418604 (21.486)

4. Secondary Outcome: Heart Rate
Description: comparison of heart rate change alfentanil vs placebo
Time Frame: Baseline and up to 30 seconds
Measure: Mean (Standard Deviation); unit: Beats per Minute
Arm/Group | Alfentanil | Placebo
Number analyzed (Participants) | 87 | 87
Beats per Minute | 37.48 (25.46) | 36.93 (25.46)

5. Secondary Outcome: Heart Rate
Description: comparison of heart rate change alfentanil vs placebo
Time Frame: 90 minutes
Population: Patients had already been discharged from the Post Anesthesia Care Unit (PACU) at 90 minutes time interval and data were not collected
Arm/Group | Alfentanil | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Maximum Heart Rate
Description: comparison of heart rate change alfentanil vs placebo
Time Frame: Baseline and up to 90 minutes
Measure: Mean (Standard Deviation); unit: Beats per Minute
Arm/Group | Alfentanil | Placebo
Number analyzed (Participants) | 87 | 87
Beats per Minute | 44.33 (24.274) | 49.66 (26.629)

7. Secondary Outcome: Minimum Heart Rate
Description: comparison of heart rate change alfentanil vs placebo
Time Frame: Baseline and up to 90 minutes
Measure: Mean (Standard Deviation); unit: Beats per Minute
Arm/Group | Alfentanil | Placebo
Number analyzed (Participants) | 87 | 87
Beats per Minute | 12.74 (14.674) | 7.08 (19.221)

8. Secondary Outcome: Doses of Antihypertensive Medication
Description: comparison of amounts of medications needed to treat blood pressure between the 2 groups
Time Frame: 90 minutes
Population: Patients had already been discharged from the PACU at 90 minutes time interval and data were not collected
Arm/Group | Alfentanil | Placebo
Number analyzed (Participants) | 0.0 | 0.0

9. Secondary Outcome: Time to Return of Spontaneous Ventilation
Description: time to return to breathing without assistance
Time Frame: up to 90 minutes
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Alfentanil | Placebo
Number analyzed (Participants) | 87 | 87
Minutes | 8.17 (2.483) | 7.25 (1.869)

10. Secondary Outcome: Total Time Subject Spent In-Room
Description: comparison of amounts time spent in-room between the 2 groups
Time Frame: up to 90 minutes
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Alfentanil | Placebo
Number analyzed (Participants) | 87 | 87
Minutes | 17.51 (4.640) | 16.43 (3.940)

11. Secondary Outcome: Severity of Headache in the Post Anesthesia Care Unit
Description: comparison between alfentanil vs placebo - Subject questionnaire with scale: 0 -10 - with 10 being the worst
Time Frame: up to 90 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alfentanil | Placebo
Number analyzed (Participants) | 87 | 87
score on a scale | 2 (2.887) | 2.467 (3.038)

12. Secondary Outcome: Satisfaction With the Anesthetic Post-procedure
Description: comparison between alfentanil vs placebo - Subject questionnaire with scale: 0-10 - with 10 being the worst
Time Frame: up to 90 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alfentanil | Placebo
Number analyzed (Participants) | 87 | 87
score on a scale | 8 (2.449) | 8.033 (2.505)

ADVERSE EVENTS:
Time Frame: 24 hours
Description: Death by suicide the day after one of their electroconvulsive therapy (ECT) procedures was completed - at which time they received Alfentanil during that ECT
Arm/Group | Alfentanil | Placebo
All-Cause Mortality (participants affected / at risk) | 1/87 | 1/87
Serious Adverse Events (participants affected / at risk) | 1/87 | 1/87
Other Adverse Events (participants affected / at risk) | 0/87 | 0/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alfentanil (N=87) | Placebo (N=87)
Suicide (Social circumstances) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alfentanil (N=87) | Placebo (N=87)
Suicide (Social circumstances) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT03359395/Prot_SAP_001.pdf
  • Informed Consent Form (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT03359395/ICF_000.pdf